CLINICAL TRIAL: NCT03717246
Title: A Sleep Hygiene Intervention to Improve Sleep Quality in Urban, Latino Middle School Children-Phase 2
Brief Title: A Sleep Hygiene Intervention to Improve Sleep Quality in Urban, Latino Middle School Children - Phase 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34HL135073 -Phase 2; 1R34HL135073 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2020-10

CONDITIONS: Sleep
Keywords: sleep hygiene; Latino Children; middle school; educational intervention
MeSH Terms: conditions — Sleep Hygiene | interventions — Child Health

STUDY DESIGN:
Intervention Model Description: 6th to 8th grade middle school students will be enrolled then randomly assigned to one of three conditions: 1) Sleep Smart Latino intervention condition , 2) child health topics education control condition; 3) a no treatment control condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleep Smart Latino (Experimental): Sleep Smart Latino is a sleep hygiene intervention culturally tailored to be consistent with the beliefs, behaviors and needs of urban Latino middle school children and families. It consists of 4 60-minute sessions delivered in a group format in an urban middle school setting, and 2 60-minute long home based sessions that involve the student and their caregiver. The intervention focuses on sleep education, including effective sleep hygiene practices, use of electronics and caffeine and their impact on sleep.
  Interventions: Behavioral: Sleep Smart Latino
- Basic Sleep Education and Child Health (Active Comparator): The basic sleep education and child health condition includes education regarding sleep hygiene , and the effects of sleep on child functioning integrated with additional child health topics such as nutrition, physical activity and safety. It consists of 4 60-minute sessions delivered in a group format in an urban middle school setting
  Interventions: Behavioral: Basic Sleep Hygiene and Child Health
- No treatment control (No Intervention): Students randomly assigned to this arm, will receive standard of care , which is no treatment and will not participate in any group sessions.

INTERVENTIONS:
Behavioral: Sleep Smart Latino — A culturally tailored group intervention aimed at improving sleep duration and quality for Latino middle school students.
  Arms: Sleep Smart Latino
Behavioral: Basic Sleep Hygiene and Child Health — A group intervention providing sleep hygiene and child health topics education to Latino middle school students.
  Arms: Basic Sleep Education and Child Health

SUMMARY:
Sleep is essential for children's daytime functioning and health. Poorer sleep hygiene can negatively affect sleep outcomes in children. Urban Latino children are at greater risk for poor sleep hygiene and poor quality sleep due to exposure to higher levels of urban and cultural stressors. This project aims to refine and test a novel school-based intervention to improve sleep hygiene and in turn, sleep quality in urban Latino middle school children. An existing sleep hygiene intervention that has been shown to improve sleep in urban children will be culturally and contextually tailored and has the potential to exert greater improvements in sleep hygiene and sleep outcomes for this high-risk group.

DETAILED DESCRIPTION:
Not sleeping long or soundly enough can lead to health problems in children, including more asthma symptoms and risk for obesity. Latino children might be especially at risk for poor sleep and worse asthma. Therefore, the goal of this study is to adapt an existing intervention called Sleep Smart for use with urban Latino middle school students. The new program will be called "Sleep Smart Latino" (SSL), the goal of which is to improve sleep quality among Latino, middle school-aged children in urban public schools. SSL will be administered by trained community members to a group of Latino middle school children who are at risk for poor sleep quality. The program will be tested in San Juan, Puerto Rico and Providence, Rhode Island.

The first aim of this project is to refine the SS intervention and intervention procedures so that they eventually can be used in a larger study of the intervention's effectiveness. Refinement will involve a) translation and cultural tailoring for Latino middle school students, b) enhancement of the parent component, and c) ensuring applicability to the urban, middle school setting in both sites (PR and RI). In-depth interviews with caregivers (N=20-25), focus groups (middle school students [N = 5], caregivers [N =5], and school staff [N = 5]), and Investigators with expertise in culturally tailored interventions will provide input.

The second aim of this application is to test the feasibility of the SSL intervention and training procedures through an Open Trial, to refine intervention modules and the training approach that will be used in the larger study. The Open Trial will include 15 adolescent participants at each study site.

The third aim of this application is to test the SSL intervention through a Pilot Randomized Control Trial to provide estimates of effect size that will be used to inform the sample size for the larger study. The RCT will include 75 adolescent participants at each study site. We expect the participants in the SSL intervention will have improvement on the following primary sleep quality outcomes (improved sleep duration and sleep efficiency) as measured by actigraphy, relative to the control conditions. Secondarily, we expect participants in SSL will show a decrease in total daily caloric intake relative to the control conditions.

This registration refers only to aims 2 and 3 of the project.

ELIGIBILITY:
Inclusion Criteria:

* specify that participants must

  1. be between the ages of 11-13,
  2. be in 6th-8th grades,
  3. reside in one of the targeted public school districts identified by zip code,
  4. attend one of the schools within these districts, and
  5. have sleep duration < 9 hours

Exclusion Criteria:

1. significant developmental delay, and/or severe psychiatric or chronic medical condition that preclude completion of study procedures or confound analyses.
2. current/prior sleep disorder diagnosis, such as sleep disordered breathing, restless leg syndrome, or periodic limb movement disorder (PLMD)

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
change in sleep duration | Assessed at baseline, immediately post intervention and 4 months post intervention
  Total sleep time: ( sleep start to sleep end) will be assessed via actigraphy data. Children will wear actigraph (Model AW4; Mini Mittler) for 2 wks at each time point. Data will be compared to diary using standard procedures
change in sleep efficiency | Assessed at baseline, immediately post intervention and 4 months post intervention
  Sleep efficiency (% epochs of sleep between sleep start and sleep end) will be assessed via actigraphy data. Children will wear actigraph (Model AW4; Mini Mittler) for 2 wks at each time point. Data will be compared to diary using standard procedures

SECONDARY OUTCOMES:
Change in total caloric intake | Assessed at baseline, immediately post intervention and 4 months post intervention
  Dietary Intake will be measured via 3 (2 week day and 1 weekend), non-consecutive 24-hour diet recalls with student at each period
Change in BMI-Z score | Assessed at baseline, immediately post intervention and 4 months post intervention
  Measures of child ht./wt. will be obtained at each period to calculate BMI z-score

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Koinis-Mitchell, PhD, Principal Investigator — Rhode Island Hospital; Glorisa Canino, PhD, Principal Investigator — University of Puerto Rico; Maria T Coutinho, PhD, Study Director — Rhode Island Hospital
Locations (2):
- Rhode Island Hospital, Providence, Rhode Island, United States
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No